CLINICAL TRIAL: NCT01165710
Title: Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF)
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Duke Clinical Research Institute (Other); Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016327; RIVAROXAFL4001 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
Keywords: Irregular heart beat
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: Patients with Atrial Fibrillation (AF) Treatment patterns of AF according to patient demographics clinical factors risk stratification and geographic regions.
  Interventions: Other: Patients with Atrial Fibrillation (AF)

INTERVENTIONS:
Other: Patients with Atrial Fibrillation (AF) — Treatment patterns of AF according to patient demographics, clinical factors, risk stratification, and geographic regions.

SUMMARY:
The ORBIT-AF registry will be a multicenter, prospective outpatient disease registry to identify "real world" treatment patterns of atrial fibrillation. The registry will describe this patient population with regards to demographics, clinical factors, risk stratification, and geographic regions. In particular, attention will be focused on the utilization, effectiveness, and safety of antithrombotic therapies in the prevention of stroke. The registry is designed to identify reasons and risk factors for non-receipt of anticoagulation (AC) therapy, as well as reasons why AF patients who are prescribed AC therapy do not take them.

DETAILED DESCRIPTION:
The ORBIT-AF registry is a multicenter prospective outpatient disease registry of patients with incident (initial diagnosis) or prevalent (existing diagnosis) atrial fibrillation (AF) that will analyze treatment patterns and outcomes in patients with AF in the US. Approximately 10,000 prospective cohort of patients will be enrolled. The registry will be a nation-wide collaboration of Health Care Providers (e.g., cardiologists, internists, primary care physicians, electrophysiologists, quality improvement personnel, office/practice managers, research coordinators, and pharmacists). This collaborative effort will be focused on the optimization of outpatient management of patients with AF. Consecutive patients who meet the eligibility criteria will be approached and educated about the registry. Patients who express interest will provide informed consent. Patients enrolled in the registry will be followed for approximately 3 years. Patient follow-up by their AF care provider will continue as scheduled according to local clinical practice. Patient Reported outcome (PRO) questionnaires will be administered to a sub-sample of approximately 1,500 patients. For patients who consent to answer PRO questionnaires, these questionnaires will be administered by the site to the patient at the baseline visit [except the baseline Anticoagulation-Related Treatment Satisfaction (ACTS)] and during their regularly scheduled follow-up visits. The baseline ACTS for incident patients will be completed and returned back to the site at least 4 weeks after starting antithrombotic therapies. The ACTS questionnaire will only be administered to patients who are taking antithrombotic therapies within the 4 weeks before a visit or newly prescribed antithrombotic therapies. Data collection will occur at 6-month intervals for a minimum of 3 years (baseline, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months). The data collection windows will be wide (3 months in either direction) in order to maximize data collection during the patients regularly scheduled follow-up with their AF care provider. Collection of Patient Reported Outcome (PRO) Questionnaires will not continue beyond the 24-month data collection interval. Atrial Fibrillation Data capture will include demographics, cardiovascular risk factors, diagnosis, type of AF (paroxysmal, persistent, permanent AF), treatment strategy (rate vs. rhythm), ablation history, cardioversions, antithrombotic therapy decisions and monitoring (INRs), concomitant medications and doses, insurance and provider information, AF quality-of-life, anticoagulation treatment satisfaction, caregiver assistance, pet ownership, comorbidities, compliance, and outcomes. Pre-defined outcomes of interest will include stroke or non-CNS (non-systemic) embolism, major adverse cardiac events, all-cause mortality, cause-specific death (sudden, non-sudden, heart failure-related), major bleeding, AF-related quality of life, anticoagulation-related treatment satisfaction, all-cause hospitalization and specific anticoagulation outcomes (e.g. time in therapeutic range and primary discontinuation of oral anticoagulation). The data generated by this registry will be used to identify real world practice, especially as it compares and relates to guidelines set forth by the American College of Cardiology, American Heart Association and European Society of Cardiology for the management of patients with AF. Observational Study - No investigational drug administered. For any patients receiving the sponsor's drug, Xarelto (rivaroxaban), under the direction of a physician, all serious adverse events and all non-serious related events will be reported to the sponsor (Janssen Scientific Affairs, LLC)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with incident (initial diagnosis) or prevalent (existing diagnosis) AF with electrocardiographic documentation
* anticipated ability to adhere to local regularly scheduled follow-up visits

Exclusion Criteria:

* Anticipated life expectancy less than 6 months
* short lasting AF secondary to a reversible condition (e.g. hyperthyroidism, pulmonary embolism, post-cardiothoracic surgery)
* Participation in a randomized trial of anticoagulation for AF at the time of enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolling physicians will include cardiologists, internists, and electrophysiologists from both academic and private practice who preferably have experience in registry participation.
Sampling Method: Non-Probability Sample
Enrollment: 10179 (Actual)
Dates: Start 2010-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is stroke or non-CNS (systemic) embolism. Key primary objective is: characterize & describe the AF patient population as a whole, with emphasis on demographics, comorbidities, and risk profiles. | 3 years

SECONDARY OUTCOMES:
The number of major adverse cardiac events. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (171):
- United States (168):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Pell City, Alabama
  - Tuscaloosa, Alabama
  - Cottonwood, Arizona
  - Tucson, Arizona
  - Fort Smith, Arkansas
  - Carlsbad, California
  - Carmichael, California
  - Corona, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Alamitos, California
  - Los Angeles, California
  - Montebello, California
  - Northridge, California
  - Orange, California
  - Oxnard, California
  - Palo Alto, California
  - Pismo Beach, California
  - Pomona, California
  - San Diego, California
  - San Ramon, California
  - Santa Rosa, California
  - Tarzana, California
  - Torrance, California
  - Tustin, California
  - Ventura, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Newark, Delaware
  - Seaford, Delaware
  - Boynton Beach, Florida
  - Coral Springs, Florida
  - Deerfield Beach, Florida
  - Fort Myers, Florida
  - Fort Walton Beach, Florida
  - Hollywood, Florida
  - Jupiter, Florida
  - Lakeland, Florida
  - Oakland Park, Florida
  - Orange Park, Florida
  - Ormond Beach, Florida
  - Port Charlotte, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Riverdale, Georgia
  - Idaho Falls, Idaho
  - Nampa, Idaho
  - Aurora, Illinois
  - Evergreen Park, Illinois
  - Melrose Park, Illinois
  - Peoria, Illinois
  - Rock Island, Illinois
  - Rockford, Illinois
  - Urbana, Illinois
  - Winfield, Illinois
  - Bloomington, Indiana
  - Evansville, Indiana
  - Hammond, Indiana
  - Indianapolis, Indiana
  - La Porte, Indiana
  - South Bend, Indiana
  - Waterloo, Iowa
  - Overland Park, Kansas
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Owensboro, Kentucky
  - Alexandria, Louisiana
  - Rockport, Maine
  - Beltsville, Maryland
  - Salisbury, Maryland
  - Biddeford, Massachusetts
  - Bay City, Michigan
  - Bridgman, Michigan
  - Commerce, Michigan
  - Grand Blanc, Michigan
  - Lansing, Michigan
  - Livonia, Michigan
  - Mount Clemens, Michigan
  - Stevensville, Michigan
  - Traverse City, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Anaconda, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Bridgewater, New Jersey
  - Elmer, New Jersey
  - Haddon Heights, New Jersey
  - Linden, New Jersey
  - Nampa, New Jersey
  - Ridgewood, New Jersey
  - Sewell, New Jersey
  - Toms River, New Jersey
  - Flushing, New York
  - Huntington, New York
  - Jamaica, New York
  - New York, New York
  - Northport, New York
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenwood, North Carolina
  - Jacksonville, North Carolina
  - Pinehurst, North Carolina
  - Raleigh, North Carolina
  - Sanford, North Carolina
  - Tabor City, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Minot, North Dakota
  - Mansfield, Ohio
  - Miamisburg, Ohio
  - Piqua, Ohio
  - Toledo, Ohio
  - Worthington, Ohio
  - Youngstown, Ohio
  - Abington, Pennsylvania
  - Beaver, Pennsylvania
  - Danville, Pennsylvania
  - Doylestown, Pennsylvania
  - Erie, Pennsylvania
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scranton, Pennsylvania
  - Spring House, Pennsylvania
  - West Reading, Pennsylvania
  - Wynnewood, Pennsylvania
  - Yardley, Pennsylvania
  - Pawtucket, Rhode Island
  - Anderson, South Carolina
  - Easley, South Carolina
  - Spartanburg, South Carolina
  - Harriman, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Beaumont, Texas
  - Corpus Christi, Texas
  - Flower Mound, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - Odessa, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - Fredericksburg, Virginia
  - Lynchburg, Virginia
  - Midlothian, Virginia
  - Roanoke, Virginia
  - Winchester, Virginia
  - Burien, Washington
  - Port Orchard, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - La Crosse, Wisconsin
  - Madison, Wisconsin
- Puerto Rico (3):
  - Hato Rey
  - Río Grande
  - San Juan

REFERENCES:
- [Derived] Fox KAA, Virdone S, Pieper KS, Bassand JP, Camm AJ, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Kayani G, Oto A, Misselwitz F, Piccini JP, Dalgaard F, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. GARFIELD-AF risk score for mortality, stroke, and bleeding within 2 years in patients with atrial fibrillation. Eur Heart J Qual Care Clin Outcomes. 2022 Mar 2;8(2):214-227. doi: 10.1093/ehjqcco/qcab028. PMID 33892489
- [Derived] Steinberg BA, Holmes DN, Pieper K, Allen LA, Chan PS, Ezekowitz MD, Freeman JV, Fonarow GC, Gersh BJ, Hylek EM, Kowey PR, Mahaffey KW, Naccarelli G, Reiffel J, Singer DE, Peterson ED, Piccini JP; ORBIT-AF (Outcomes Registry for Better Informed Treatment of Atrial Fibrillation) Investigators and Patients. Factors Associated With Large Improvements in Health-Related Quality of Life in Patients With Atrial Fibrillation: Results From ORBIT-AF. Circ Arrhythm Electrophysiol. 2020 May;13(5):e007775. doi: 10.1161/CIRCEP.119.007775. Epub 2020 Apr 16. PMID 32298144
- [Derived] Holmes DN, Piccini JP, Allen LA, Fonarow GC, Gersh BJ, Kowey PR, O'Brien EC, Reiffel JA, Naccarelli GV, Ezekowitz MD, Chan PS, Singer DE, Spertus JA, Peterson ED, Thomas L. Defining Clinically Important Difference in the Atrial Fibrillation Effect on Quality-of-Life Score. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005358. doi: 10.1161/CIRCOUTCOMES.118.005358. PMID 31092022
- [Derived] Thind M, Holmes DN, Badri M, Pieper KS, Singh A, Blanco RG, Steinberg BA, Fonarow GC, Gersh BJ, Mahaffey KW, Peterson ED, Reiffel JA, Piccini JP, Kowey PR; ORBIT-AF Investigators and Patients. Embolic and Other Adverse Outcomes in Symptomatic Versus Asymptomatic Patients With Atrial Fibrillation (from the ORBIT-AF Registry). Am J Cardiol. 2018 Nov 15;122(10):1677-1683. doi: 10.1016/j.amjcard.2018.07.045. Epub 2018 Aug 20. PMID 30227964
- [Derived] Durheim MT, Holmes DN, Blanco RG, Allen LA, Chan PS, Freeman JV, Fonarow GC, Go AS, Hylek EM, Mahaffey KW, Pokorney SD, Reiffel JA, Singer DE, Peterson ED, Piccini JP. Characteristics and outcomes of adults with chronic obstructive pulmonary disease and atrial fibrillation. Heart. 2018 Nov;104(22):1850-1858. doi: 10.1136/heartjnl-2017-312735. Epub 2018 Jun 6. PMID 29875139
- [Derived] O'Brien EC, Holmes DN, Thomas LE, Fonarow GC, Allen LA, Gersh BJ, Kowey PR, Singer DE, Ezekowitz MD, Naccarelli GV, Ansell JE, Chan PS, Mahaffey KW, Go AS, Freeman JV, Reiffel JA, Peterson ED, Piccini JP, Hylek EM. Prognostic Significance of Nuisance Bleeding in Anticoagulated Patients With Atrial Fibrillation. Circulation. 2018 Aug 28;138(9):889-897. doi: 10.1161/CIRCULATIONAHA.117.031354. PMID 29678813
- [Derived] Fox KAA, Lucas JE, Pieper KS, Bassand JP, Camm AJ, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Hacke W, Kayani G, Oto A, Mantovani LG, Misselwitz F, Piccini JP, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. Improved risk stratification of patients with atrial fibrillation: an integrated GARFIELD-AF tool for the prediction of mortality, stroke and bleed in patients with and without anticoagulation. BMJ Open. 2017 Dec 21;7(12):e017157. doi: 10.1136/bmjopen-2017-017157. PMID 29273652
- [Derived] Piccini JP, Simon DN, Steinberg BA, Thomas L, Allen LA, Fonarow GC, Gersh B, Hylek E, Kowey PR, Reiffel JA, Naccarelli GV, Chan PS, Spertus JA, Peterson ED; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Investigators and Patients. Differences in Clinical and Functional Outcomes of Atrial Fibrillation in Women and Men: Two-Year Results From the ORBIT-AF Registry. JAMA Cardiol. 2016 Jun 1;1(3):282-91. doi: 10.1001/jamacardio.2016.0529. PMID 27438106
- [Derived] Golwala H, Jackson LR 2nd, Simon DN, Piccini JP, Gersh B, Go AS, Hylek EM, Kowey PR, Mahaffey KW, Thomas L, Fonarow GC, Peterson ED, Thomas KL; Outcomes Registry for Better Informed Treatment for Atrial Fibrillation (ORBIT-AF) Registry. Racial/ethnic differences in atrial fibrillation symptoms, treatment patterns, and outcomes: Insights from Outcomes Registry for Better Informed Treatment for Atrial Fibrillation Registry. Am Heart J. 2016 Apr;174:29-36. doi: 10.1016/j.ahj.2015.10.028. Epub 2015 Dec 30. PMID 26995367
- [Derived] Jackson LR 2nd, Kim SH, Piccini JP Sr, Gersh BJ, Naccarelli GV, Reiffel JA, Freeman J, Thomas L, Chang P, Fonarow GC, Go AS, Mahaffey KW, Peterson ED, Kowey PR. Sinus Node Dysfunction Is Associated With Higher Symptom Burden and Increased Comorbid Illness: Results From the ORBIT-AF Registry. Clin Cardiol. 2016 Feb;39(2):119-25. doi: 10.1002/clc.22504. Epub 2015 Dec 31. PMID 26720750
- [Derived] Steinberg BA, Kim S, Thomas L, Fonarow GC, Gersh BJ, Holmqvist F, Hylek E, Kowey PR, Mahaffey KW, Naccarelli G, Reiffel JA, Chang P, Peterson ED, Piccini JP; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Investigators and Patients. Increased Heart Rate Is Associated With Higher Mortality in Patients With Atrial Fibrillation (AF): Results From the Outcomes Registry for Better Informed Treatment of AF (ORBIT-AF). J Am Heart Assoc. 2015 Sep 14;4(9):e002031. doi: 10.1161/JAHA.115.002031. PMID 26370445
- [Derived] Holmqvist F, Simon D, Steinberg BA, Hong SJ, Kowey PR, Reiffel JA, Naccarelli GV, Chang P, Gersh BJ, Peterson ED, Piccini JP; ORBIT-AF Investigators. Catheter Ablation of Atrial Fibrillation in U.S. Community Practice--Results From Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF). J Am Heart Assoc. 2015 May 21;4(5):e001901. doi: 10.1161/JAHA.115.001901. PMID 25999401
- [Derived] Holmqvist F, Guan N, Zhu Z, Kowey PR, Allen LA, Fonarow GC, Hylek EM, Mahaffey KW, Freeman JV, Chang P, Holmes DN, Peterson ED, Piccini JP, Gersh BJ; ORBIT-AF Investigators. Impact of obstructive sleep apnea and continuous positive airway pressure therapy on outcomes in patients with atrial fibrillation-Results from the Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF). Am Heart J. 2015 May;169(5):647-654.e2. doi: 10.1016/j.ahj.2014.12.024. Epub 2015 Feb 7. PMID 25965712
- [Derived] Steinberg BA, Peterson ED, Kim S, Thomas L, Gersh BJ, Fonarow GC, Kowey PR, Mahaffey KW, Sherwood MW, Chang P, Piccini JP, Ansell J; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation Investigators and Patients. Use and outcomes associated with bridging during anticoagulation interruptions in patients with atrial fibrillation: findings from the Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF). Circulation. 2015 Feb 3;131(5):488-94. doi: 10.1161/CIRCULATIONAHA.114.011777. Epub 2014 Dec 12. PMID 25499873
- [Derived] Steinberg BA, Kim S, Fonarow GC, Thomas L, Ansell J, Kowey PR, Mahaffey KW, Gersh BJ, Hylek E, Naccarelli G, Go AS, Reiffel J, Chang P, Peterson ED, Piccini JP. Drivers of hospitalization for patients with atrial fibrillation: Results from the Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF). Am Heart J. 2014 May;167(5):735-42.e2. doi: 10.1016/j.ahj.2014.02.003. Epub 2014 Feb 17. PMID 24766985
- [Derived] Steinberg BA, Kim S, Thomas L, Fonarow GC, Hylek E, Ansell J, Go AS, Chang P, Kowey P, Gersh BJ, Mahaffey KW, Singer DE, Piccini JP, Peterson ED; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Investigators and Patients. Lack of concordance between empirical scores and physician assessments of stroke and bleeding risk in atrial fibrillation: results from the Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) registry. Circulation. 2014 May 20;129(20):2005-12. doi: 10.1161/CIRCULATIONAHA.114.008643. Epub 2014 Mar 29. PMID 24682387
- [Derived] Steinberg BA, Holmes DN, Piccini JP, Ansell J, Chang P, Fonarow GC, Gersh B, Mahaffey KW, Kowey PR, Ezekowitz MD, Singer DE, Thomas L, Peterson ED, Hylek EM; Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Investigators and Patients. Early adoption of dabigatran and its dosing in US patients with atrial fibrillation: results from the outcomes registry for better informed treatment of atrial fibrillation. J Am Heart Assoc. 2013 Nov 25;2(6):e000535. doi: 10.1161/JAHA.113.000535. PMID 24275632
- [Derived] Steinberg BA, Kim S, Piccini JP, Fonarow GC, Lopes RD, Thomas L, Ezekowitz MD, Ansell J, Kowey P, Singer DE, Gersh B, Mahaffey KW, Hylek E, Go AS, Chang P, Peterson ED; ORBIT-AF Investigators and Patients. Use and associated risks of concomitant aspirin therapy with oral anticoagulation in patients with atrial fibrillation: insights from the Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT-AF) Registry. Circulation. 2013 Aug 13;128(7):721-8. doi: 10.1161/CIRCULATIONAHA.113.002927. Epub 2013 Jul 16. PMID 23861512
- [Derived] Piccini JP, Fraulo ES, Ansell JE, Fonarow GC, Gersh BJ, Go AS, Hylek EM, Kowey PR, Mahaffey KW, Thomas LE, Kong MH, Lopes RD, Mills RM, Peterson ED. Outcomes registry for better informed treatment of atrial fibrillation: rationale and design of ORBIT-AF. Am Heart J. 2011 Oct;162(4):606-612.e1. doi: 10.1016/j.ahj.2011.07.001. PMID 21982650